CLINICAL TRIAL: NCT03834792
Title: Adverse Long-term Consequences of Sleep Disordered Breathing: Using the Ottawa Hospital Sleep Database in Predictive Model Development and Validation.
Brief Title: Adverse Long-term Consequences of Sleep Disordered Breathing: The Ottawa Hospital (TOH) Sleep Database
Status: Active, not recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other); University of Toronto (Other); University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 20170591-01H
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Polysomnography; Sleep Apnea Syndromes; Risk Factors; Prognosis; Restless Legs Syndrome; Periodic Limb Movement Sleep Disorder; Sleep Arousal Disorders; Opioid Use
Keywords: Sleep disorders; Health outcomes; Predictive model; Health care utilization; Validation
MeSH Terms: conditions — Sleep Apnea Syndromes; Restless Legs Syndrome; Sleep Arousal Disorders; Sleep Wake Disorders; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention but exposure — Different sleep disorders will be considered as an exposure. The data elements included in the database: demographics, date of the sleep study, study type, all available polysomnography indices, symptoms, sleep schedule, comorbidities, medications, social history, electrocardiography, positive airway pressure treatment related variables.

SUMMARY:
The primary purpose of the proposed study is to validate our previously developed predictive model for adults with obstructive sleep apnea using (i) clinical data from multiple large academic centers, (ii) a longer follow-up period, and (iii) an extended definition of outcomes of interest.

The TOH sleep database was created as a part of the project: "Validation of provincial health administrative data algorithms to identify patients with obstructive sleep apnea (OSA): Feasibility project". Protocol ID: 20170591-01H (AMENDMENT APPROVED on December 19, 2018) to be used for future clinical, research, educational and quality improvement purposes.

DETAILED DESCRIPTION:
The primary purpose of the proposed study is to validate the previously developed predictive model by the investigators for adults with obstructive sleep apnea using (i) clinical data from multiple large academic centers, (ii) a longer follow-up period, and (iii) an extended definition of outcomes of interest.

From clinical and quality improvement perspective the TOH database will be used for description, evaluation, monitoring and/or educational purposes. For example, using this database the investigators will be able (i) to describe characteristics of individuals who underwent a diagnostic sleep study at the TOH between 2015 and 2017 to understand better clinical and health care utilization needs as well as to educate sleep fellows and technologists; and (ii) to evaluate the quality of the triaging process in the sleep clinic. This database will be used to: (i) examine risk factors for long-term adverse health consequences (e.g. cardio-vascular diseases, diabetes, depression, dementia, depression and cancer) among individuals referred for diagnostic sleep testing in order to identify high risk groups that are potential targets for education and treatment, (ii) develop health interventions in order to improve the quality of care and management strategies available for adults with chronic diseases that are comorbid with obstructive airway diseases and sleep-related disorders, (iii) evaluate the cost-effectiveness of the developed health interventions, e.g. screening for obstructive sleep apnea (OSA), evaluation of home versus laboratory-based diagnosis of OSA, and education strategies, (iv) develop key messages for different stakeholder groups (health care providers, patients and their relatives, provincial sleep and lung associations, public health managers, the respiratory vendor among others) related to diagnosis, education and treatment of patients with respiratory and sleep-related problems.

ELIGIBILITY:
Inclusion criteria:

• All adults who underwent a diagnostic sleep study in the TOH Sleep Center from Apr 2015 to April 2017

Exclusion criteria:

* Uninsured individuals
* Individuals who did not agree for their data to be linked to the ICES
* Individuals who underwent split-night sleep studies

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Please see above
Sampling Method: Non-Probability Sample
Enrollment: 5155 (Estimated)
Dates: Start 2018-12-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Long-term adverse health consequences | Through study completion, up to 10 years
  The primary outcome will be time from the index date (diagnostic sleep study) to the composite outcome of interest which include: cardio-vascular diseases, diabetes, depression, dementia, and cancer as well as chronic lung diseases and all-cause mortality. Conditions of interested will be defined from provincial health administrative data using validated algorithms that have utilized ICD-9 and ICD-10 codes as well as billing codes for outpatients visits, and procedural codes. Please see ICES Data Dictionary for details: https://www.ices.on.ca/Data-and-Privacy/ICES-data/Data-dictionary.

SECONDARY OUTCOMES:
Health care utilization | Through study completion, up to 10 years
  All-cause mortality, all-cause hospitalizations, emergency department visits and associated costs will be defined from provincial health administrative data. Registered Persons Database will be used to define mortality. Hospitalizations and emergency department visits will be defined using: Discharge Abstract Database (all hospital admission and discharge data), National Ambulatory Care Reporting System (emergency department visits). Please see ICES Data Dictionary for details: https://www.ices.on.ca/Data-and-Privacy/ICES-data/Data-dictionary. Total healthcare expenditures will be calculated using the ICES person-level health utilization costing algorithms.
Motor vehicle crashes | Through study completion, up to 10 years
  Different definitions of motor vehicle crashes will be considered. Motor vehicle crashes requiring hospital or emergency department visit: the investigators will identify traffic emergencies characterized as a crash using the International Classification of Diseases codes 10th Revision (V20-V69). The investigators will include emergency department visits involving crashes in which the patient was the driver of the motor vehicle and exclude emergency department visits involving crashes in which the patient was a passenger or pedestrian.

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Kendzerska, MD, PhD, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided yet if IPD will be available to other researchers.

REFERENCES:
- [Derived] Kendzerska T, Murray BJ, Gershon AS, Povitz M, McIsaac DI, Bryson GL, Talarico R, Hilton J, Malhotra A, Leung RS, Boulos MI. Polysomnographic Assessment of Sleep Disturbances in Cancer Development: A Historical Multicenter Clinical Cohort Study. Chest. 2023 Aug;164(2):517-530. doi: 10.1016/j.chest.2023.03.006. Epub 2023 Mar 11. PMID 36907376